CLINICAL TRIAL: NCT00592085
Title: Combined Treatment for Tobacco and Alcohol Use
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No patients registered; study terminated.
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2007-0111
Record Dates: First submitted 2007-12-27; First posted 2008-01-11 (Estimated); Last update posted 2016-07-20 (Estimated); Status verified 2009-09

CONDITIONS: Smoking Cessation
Keywords: Tobacco Use; Smoking; Alcohol Use; Smoking Cessation
MeSH Terms: conditions — Smoking Cessation; Tobacco Use; Smoking; Alcohol Drinking | interventions — Surveys and Questionnaires; Ethanol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Relapse Prevention Counseling (Active Comparator): Motivational Relapse Counseling: 6 counseling calls over two weeks accompanied by questionnaires
  Interventions: Behavioral: Questionnaires; Behavioral: Motivational Relapse Prevention Counseling
- Relapse Prevention + Alcohol Counseling (Active Comparator): Motivational Relapse Prevention Plus Alcohol Risk Reduction Counseling: 6 counseling calls over two weeks for both smoking cessation and at-risk alcohol use accompanied by questionnaires
  Interventions: Behavioral: Questionnaires; Behavioral: Relapse Plus Alcohol Risk Reduction Counseling

INTERVENTIONS:
Behavioral: Questionnaires — Participants will use a computer to complete a series of questionnaires.
Behavioral: Motivational Relapse Prevention Counseling — Total of 6 counseling calls for Smoking Relapse: First counseling call will be to set up your quit date; then 5 additional counseling calls within 12 weeks after enrollment, each 20 to 30 minutes to complete.
  Arms: Relapse Prevention Counseling
Behavioral: Relapse Plus Alcohol Risk Reduction Counseling — Total of 6 counseling calls for both Smoking Relapse and Alcohol Risk: First counseling call will be to set up your quit date; then 5 additional counseling calls within 12 weeks after enrollment, each 20 to 30 minutes to complete.
  Arms: Relapse Prevention + Alcohol Counseling

SUMMARY:
The specific aims are to:

* Develop a "Motivational Relapse Prevention Plus Alcohol Risk Reduction" (MRP+) approach to simultaneously treating both smoking and "at-risk" alcohol use among smokers attempting to quit smoking.
* Estimate the effect size for MRP+ relative to Motivational Relapse Prevention without a focus on alcohol (MRP) with respect to alcohol at-risk behaviors. The estimated effect size will be utilized to help guide sample size estimates for a potential clinical trial.

DETAILED DESCRIPTION:
Study Participation If you agree to take part in this study, you will come to M. D. Anderson and use a computer to complete a series of questionnaires. You will be asked questions about your living situation, mood, depression, anxiety, appetite, smoking and alcohol use habits, social status, finances, job, physical activity, and support from family and/or friends. These questionnaires may take a total of about 1 hour to complete.

After completing the questionnaires, you will be randomly assigned (as in the toss of a coin) to one of two groups. One group will receive counseling (called motivational relapse prevention counseling), which will focus on smoking cessation. The other group will also receive counseling (called motivational relapse prevention plus alcohol risk reduction counseling), which will focus on smoking cessation as well but will also include discussion about at-risk alcohol use. Both groups will receive reading materials related to smoking cessation. The motivational relapse prevention plus alcohol risk reduction group will also receive reading materials related to alcohol use.

You will receive a total of 6 counseling calls during this study. Your first counseling call will be to set up your quit date. You will then have 5 additional counseling calls within the 12 weeks after your enrollment in the study. The timing of these calls will be determined between you and your counselor. Depending on which group you are in, you will be counseled on strategies for quitting smoking and/or decreasing alcohol use to help decrease your risk of cancer. These calls will take about 20 to 30 minutes each to complete. You will be asked to provide contact information for friends and/or relatives. The research staff will contact them only if you are unable to be contacted after multiple attempts.

Final Visit At Week 12, you will be requested to return to M. D. Anderson to complete the last computerized series of questionnaires.

Your counseling calls will be tape recorded so researchers can make sure that correct procedures are being followed. Only the study staff will be allowed to listen to these tapes. Your identity will be kept secure and confidential. These tapes will be erased when this study has ended.

Study Length Your participation in this study will be over after the evaluation visit at Week 12.

ELIGIBILITY:
Inclusion Criteria:

* Current daily smoker who averages 5 or more cigarettes/day.
* Exhibit at least one of the following criteria for at-risk drinking: a) an average of > or equal to 2 alcoholic beverages/day during the past 30 days for men or > or equal to 1 drink/day for women, OR b) two or more occasions of consuming > or equal to 5 alcoholic beverages during the past 30 days for men or > or equal to 4 drinks for women, OR c) driving after consuming > or equal to 3 drinks in the past 30 days,
* Age 18 or above
* Motivated to quit smoking in the next 30 days
* Viable (working) telephone number and home address
* No other household member enrolled in this protocol
* Score equal to or less than 15 on the Alcohol Use Disorders Identification Test (AUDIT) measure.
* Must be able to speak English.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-12; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Overall at-risk drinking status | Baseline and Week 12
  At-risk drinking, defined by National Institute on Alcohol Abuse and Alcoholism, refers to a constellation of alcohol use behaviors that increase risk for physical and psychosocial problems including (a) an average of > 2 alcoholic beverages/day during the past 30 days for men or >1 drink/day for women, OR (b) two or more occasions of consuming > 5 alcoholic beverages during the past 30 days for men or >4 drinks for women, OR (c) driving after consuming >3 drinks in the past 30 days.

SECONDARY OUTCOMES:
Effectiveness of certain type of telephone counseling ability to help participants decrease both their smoking and at-risk alcohol use as measured by Smoking Cessation and At-Risk Drinking Evaulation | Up to 3 months for baseline and repeat assessments at 12 weeks
  Effectiveness evaluated using descriptive data from questionnaires to evaluate theoretically- and empirically-based "Motivational Relapse Prevention Plus Alcohol Risk Reduction" (MRP+) approach for simultaneously intervening on both smoking and at risk alcohol use. Evaluation through questionnaire results, smoking cessation and overall at-risk drinking status, a dichotomous variable defined previously.

CONTACTS AND LOCATIONS:
Overall Officials: David Wetter, PHD, MS, BA, Principal Investigator — M.D. Anderson Cancer Center

REFERENCES:
- See also: MD Anderson Cancer Center website — http://www.mdanderson.org